CLINICAL TRIAL: NCT06017531
Title: Ultrasonographic Characterization of Parametrial Lesions in Deep Endometriosis: A Diagnostic-Accuracy Study (ULTRA-PARAMETRENDO III)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center, prospective diagnostic-accuracy study. All women who will undergo surgery for DE after preoperative ultrasound for six consecutive months will be included. Anamnestic and preoperative (physical objective and ultrasonographic) data of these patients will be collected. Surgical and pathological data will be analyzed to confirm the presence of parametrial DE.

DETAILED DESCRIPTION:
This is a single-center, prospective diagnostic-accuracy study. All women who will undergo surgery for DE after preoperative ultrasound for six consecutive months will be included. Anamnestic and preoperative (physical objective and ultrasonographic) data of these patients will be collected. Surgical and pathological data will be analyzed to confirm the presence of parametrial DE.

All the study procedures are done according to our clinical practice. Demographic and ultrasonographic data will be collected from the preoperative evaluation, which is routinely done at our institution by four ultrasonographic expert in diagnosing deep endometriosis. Surgical and pathological data will be collected during surgical procedures and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of DE, for which a preoperative transvaginal ultrasonographic assessment and laparoscopic surgical approach will be indicated;
* age > or equal to 18 years
* informed consent for the participation in the study and for personal data treatment.

Exclusion Criteria:

* previous surgical diagnosis of parametrial DE;
* previous radiological diagnosis of parametrial DE including techniques used to diagnose DE (such as magnetic resonance [MRI], computed tomography-based virtual colonoscopy [CTC] or double-contrast barium enema);
* previous bilateral ovariectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who will undergo surgery for DE after preoperative ultrasound for six consecutive months will be included.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Preoperative exam, surgical and/or histological confirmation
  Diagnostic accuracy of transvaginal ultrasound for detecting the intraoperative presence of parametrial DE with surgical and/or histological confirmation.
Sensitivity | Preoperative exam, surgical and/or histological confirmation
  Sensitivity of transvaginal ultrasound for detecting the intraoperative presence of parametrial DE with surgical and/or histological confirmation.
Specificity | Preoperative exam, surgical and/or histological confirmation
  Specificity of transvaginal ultrasound for detecting the intraoperative presence of parametrial DE with surgical and/or histological confirmation.
positive predictive value | Preoperative exam, surgical and/or histological confirmation
  of transvaginal ultrasound for detecting the intraoperative presence of parametrial DE with surgical and/or histological confirmation.
negative predictive value | Preoperative exam, surgical and/or histological confirmation
  of transvaginal ultrasound for detecting the intraoperative presence of parametrial DE with surgical and/or histological confirmation.
Positive likelihood ratio | Preoperative exam, surgical and/or histological confirmation
  Positive likelihood ratio of transvaginal ultrasound for detecting the intraoperative presence of parametrial DE with surgical and/or histological confirmation.
Negative likelihood ratio | Preoperative exam, surgical and/or histological confirmation
  Negative likelihood ratio of transvaginal ultrasound for detecting the intraoperative presence of parametrial DE with surgical and/or histological confirmation.

SECONDARY OUTCOMES:
Characteristics of parametrial DE | Preoperative exam
  Characteristics of parametrial DE (parametrial localizations, size, margins, echogenicity) evaluated at preoperative ultrasound
Parametrial DE in the three different parametrial areas (posterior, lateral, and anterior parametrium) | Preoperative exam, surgical and/or histological confirmation
  Diagnostic accuracy, sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, and negative likelihood ratio of transvaginal ultrasound for distinguishing the intraoperative presence of parametrial DE in the three different parametrial areas (posterior, lateral, and anterior parametrium) with surgical and/or histological confirmation.
Infiltration of parametrial DE nodules | Preoperative exam, surgical and/or histological confirmation
  Diagnostic accuracy, sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, and negative likelihood ratio of transvaginal ultrasound for detecting the intraoperative infiltration of parametrial DE nodules in other pelvic structures (i.e. rectosigmoid, uterosacral ligaments) with surgical and/or histological confirmation
Other DE nodules and indirect DE signs | Preoperative exam
  Prevalence of other DE nodules and indirect DE signs in patients in the case of evidence of parametrial DE at preoperative ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria di Negrar, Negrar, Verona, Italy

REFERENCES:
- [Derived] Barra F, Zorzi C, Albanese M, De Mitri P, Stepniewska A, Roviglione G, Giani M, Albertini G, Ferrero S, Ceccaroni M. Ultrasonographic characterization of parametrial endometriosis: a prospective study. Fertil Steril. 2024 Jul;122(1):150-161. doi: 10.1016/j.fertnstert.2024.02.031. Epub 2024 Feb 19. PMID 38382700